CLINICAL TRIAL: NCT07296874
Title: Acute Effects of Cannabis on Cognition and Affect
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington State University (Other)
Responsible Party: Principal Investigator, Ryan Mclaughlin, Associate Professor, Washington State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 25-0421
Record Dates: First submitted 2025-12-03; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cannabis Use
Keywords: Cannabis; THC; Executive functioning; Stress reactivity; Affect
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, crossover clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and the research assistants who administer the cognitive assessments (and other outcomes) will be blinded to the drug condition. The PI (Dr. McLaughlin) will be unblinded and will handle the drug, including weighing and pre-loading it into the Volcano vaporizer prior to each testing session. Additionally, the PI (Dr. McLaughlin or Dr. Cuttler) who supervises the vaping session will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- THC -> Placebo (Experimental): Participants will inhale vapor from .17 grams of cannabis containing 11.86% THC (20mg THC total) during the first session. They will inhale vapor from a placebo product during the second session.
  Interventions: Drug: THC 20mg; Drug: Placebo
- Placebo -> THC (Experimental): Participants will inhale vapor from a placebo product during the first session. They will inhale vapor from .17 grams of cannabis containing 11.86% THC (20mg THC total) during the second session.
  Interventions: Drug: THC 20mg; Drug: Placebo

INTERVENTIONS:
Drug: THC 20mg — 20 mg THC delivered by vaporizing 0.17 g of 11.86% THC cannabis flower obtained from NIDA, using a Volcano vaporizer.
Drug: Placebo — Placebo obtained from NIDA and vaporized using a Volcano vaporizer.

SUMMARY:
This study will examine how a moderate dose of THC affects mood, stress responses, and cognitive functioning in regular cannabis users. The study uses a double-blind, placebo-controlled, crossover design, meaning each participant will complete two sessions. Specifically, each participant will be given active cannabis (20 mg THC) in one session, and placebo in the other session. The order will be randomized across participants, so half will receive cannabis first, and the other half will receive placebo first.

Ninety adults who use cannabis at least weekly will be recruited from the local community. After an online screening survey, eligible participants will attend a laboratory visit where the participants will provide informed consent and complete saliva and urine drug tests to confirm recent abstinence from cannabis and absence of other drugs. Participants who pass screening will complete baseline questionnaires of cannabis use patterns, depression, anxiety, ADHD symptoms, emotion regulation, affect, and demographic information.

Cannabis and placebo materials (obtained from NIDA) will be vaporized using a Volcano vaporizer device. Participants will inhale the vapor under supervision, and neither the participant nor the researcher assessing outcomes will know which product is administered. After vaping, participants will complete repeated mood ratings, saliva samples, and a battery of cognitive tests assessing executive functions like planning, inhibition, working memory, and cognitive flexibility.

Participants will also complete a standardized stress challenge (the Maastricht Acute Stress Test), which involves repeated trials of placing their hand in cold water and doing challenging mental math, followed by additional mood ratings and saliva samples. The participants will then watch a nature video and report their feelings of awe and affect.

At the end of each session, participants will remain in a supervised room with entertainment and snacks until at least four hours have passed since vaping and the participants report feeling sober. The participants will then return for a second session with the opposite study condition (THC or placebo) one week later. Both sessions follow the same procedures. Participants are fully debriefed after completing the study.

DETAILED DESCRIPTION:
Design: The investigators will address the research questions using a double-blind, placebo-controlled, crossover design.

Cannabis Procurement, Storage, and Transport: Cannabis will be obtained from the National Institute on Drug Abuse (NIDA). The investigators will obtain cannabis containing 11.86% THC (barrel #1592). Our plan for dosing considers potency (grams of flower x 1000 x %THC = mg THC), so participants in the 20 mg THC condition will be administered .17g of 11.86% THC cannabis flower. The placebo will also be obtained from NIDA.

Cannabis will be stored in the PI's secure cannabis storage facilities in the Veterinary and Biomedical Research (VBRB) building. A maximum of 24 hours before a scheduled testing session, an individual authorized by the DEA will transport a small amount of cannabis or placebo (corresponding to 20 mg THC) from the secure VBRB storage facilities to the psychology building, where participants will vape the cannabis. The product will be stored in the chamber of a Volcano Vaporizer in a locked room.

Recruitment: A total of 90 cannabis users will be recruited from Pullman and the neighboring communities. Advertisements will be placed in local cannabis dispensaries and on social media (e.g., Facebook Free & For Sale, Reddit, Instagram). The investigators will also email chronic cannabis users who have participated in our former cannabis studies (and have indicated willingness to be contacted with invitations for subsequent studies) to invite them to participate. These advertisements and emails will include a link to an online Qualtrics survey used to determine eligibility. This survey will be used to screen for serious psychiatric conditions (psychosis, bipolar I, panic disorder), a family history of psychosis, neurological disorders, chronic medical conditions (e.g., heart disease, diabetes, Reynaud's disease), a body mass index (BMI) exceeding 34, learning disabilities, intellectual disabilities, history of multiple concussions or head injury that may impact cognition, pregnancy or lactation, and history of adverse experiences with cannabis (psychosis, panic attacks), use of illicit drugs in the past 6 months, heavy alcohol use (>4 drinks, >4 times/week), and smoking/nicotine use. Eligible participants will need to have used cannabis at least once a week for at least one year, the participants will need to indicate that they typically inhale cannabis, and be willing to abstain from using any cannabis on the day of their scheduled testing session (minimum of 8 hours of abstinence). This survey will be used to obtain contact information from interested and eligible candidates. Ineligible participants will not be given the opportunity to enter their contact information, so sensitive information will only be collected from anonymous individuals. Eligible candidates will be contacted using the contact information provided, and the testing session will be scheduled. Participants will be instructed not to use any cannabis on the day of the testing session (from midnight onward).

Consent & Drug Screen: Participants will meet the research assistant in The Health & Cognition (THC) lab in the Department of Psychology at WSU. After obtaining written informed consent, participants will be asked when they last ate and drank (anything but water) and when they last used cannabis. Participants who report using cannabis that day will be rescheduled and will be reminded that they must abstain from any cannabis use on the day of the testing session. To further verify abstinence from cannabis on the day of the testing session, the participants will be asked to complete a THC saliva test. The participants will then be asked to complete a 12-panel urine drug test to ensure the participants test negative for illicit drugs. Participants who test positive for illicit drugs are not eligible and will not be permitted to complete the study.

Survey and Baseline Assessments: Participants who pass the drug test (test negative for illicit drugs), will be asked to put on an Embrace medical-grade wristband, the research assistant (RA) will place a Muse S Athena EEG headband on them, and the participants will be asked to provide a small saliva sample (from which cortisol will be extracted) by chewing on a Salivette for 1 minute and then spitting the saturated Salivette in a sterile tube. The participants will then rate how high they feel using a scale from 0 = "not high at all" to 10 = "extremely high." Next, the participants will complete standardized, valid, and reliable measures of their cannabis consumption patterns (Daily Sessions, Frequency, Age of Onset, and Quantity of Cannabis Use Inventory), depression (Center for Epidemiologic Studies Depression Scale [CES-D]), anxiety (Beck Anxiety Inventory [BAI]), ADHD symptoms (Barkley Adult ADHD Rating Scale - IV), emotion regulation (Difficulties in Emotion Regulation Scale [DERS]), affect (Daniels Five-Factor Measure of Affective Well-Being [D-FAW]), and demographic information. The information from this survey will be used to characterize the sample, determine covariates that should be controlled for in analyses, and examine the potential moderating effects of depression/anxiety/emotion regulation on cannabis induced changes in mood, anxiety, and affect. Participants will then complete the Wechsler Test of Adult Reading as an index of verbal IQ.

Drug Administration: Once the baseline assessments have been obtained, the researcher will bring the participant to the vaping room for their vaping session. This is a secluded room (none of the neighboring rooms are currently in use by people) in the basement of the building with a functioning fume hood. The researcher will position the Volcano Vaporizer pre-loaded with cannabis containing 20 mg of THC or placebo (the researcher and participant will be blind to the product) near the participant. The researcher will turn the vaporizer on and will wait until it heats up to 210 degrees Celsius. This temperature is ideal as it is not hot enough for the plant material to burn, so many of the toxins associated with smoking are not released. The researcher will set up a Zoom videoconferencing session on an iPad/computer and will text one of the principal investigators (PIs) to join the Zoom call. Importantly, this Zoom session will NOT be recorded. The RA will then go to an adjacent room and wait until the cannabis session is complete to aid with their blinding to the drug condition. Once one of the PIs joins the Zoom call, the investigators will instruct the participant to begin inhaling the vapor and exhaling into a "sploofy" carbon filter. The participants will be asked to try to inhale for a minimum of 2 seconds, and hold for 2 seconds, before exhaling into the sploofy. The PI will count the total number of puffs the participant inhales and will time the duration of their inhalations and holds. Once the participant has inhaled 30 puffs, they will be asked to exhale into the air and to look to see if there is any visible vapor. If the participants see visible vapor, they will continue to take more puffs and exhale into the sploofy. Every 5-10 puffs, the participants will exhale into the air to see if they notice any vapor. This will continue until the participants don't see any vapor. The PI will ask the participant to rate how high they feel using a scale from 0 = "not high at all" to 10 = "extremely high." The participants will also rate the level of good drug effects they are experiencing and their liking of those drug effects using similar 0 to 10 scales. The PI will text the RA when the vaping session is complete, and the RA will return, clean the mouthpiece with rubbing alcohol, put the Volcano Vaporizer away, and turn on the fume hood. The RA will then bring the participant back to the original lab room to complete the cognitive tests.

Cognitive Tests: Participants will be asked to rate their affect using the D-FAW and then be asked to provide another saliva sample (from which cortisol will be extracted). Participants will be asked to complete cognitive tests of planning, inhibition, task switching, and working memory, including tests of prospective memory, the N-back, digit span backwards, tower test, zoo maps test, Stroop test, oddball task, flanker task, Wisconsin card sorting test, and verbal fluency category switching tests.

Stress Challenge: Participants will then complete the Maastricht Acute Stress Test. This test includes a physical stress challenge, a cognitive challenge, and elements of unpredictability and uncontrollability. The investigators have slightly modified the task to remove the minor deception that the participants are being video-recorded during the task. Participants will be asked to place their hand in a cooler of cold water (1-3 °C) for a predetermined yet undisclosed length of time (not to exceed 90s). Immediately after each immersion trial, participants will be instructed to complete a mental arithmetic task (counting backwards from 2043 by 17s). Each time the participants make a mistake, they will be given negative feedback and instructed to start over. Once the computer signals the start of their next hand immersion trial, the participants will stop the mental arithmetic and place their hand back in the water. The participants will continue to alternate between immersion and mental arithmetic until completing 5 immersion trials of varying duration (that never exceed 90 s) and four arithmetic trials of varying durations. Immediately before and after the stress test, the participants will provide saliva samples (from which cortisol, oxytocin, and inflammatory cytokines will be extracted), and will rate their affect using the D-FAW, and the strength of their subjective high, good drug effects and liking of the drug effects using 0 (not at all) to 10 (extremely) scales on an iPad.

Nature Video and AWE: Participants will then be brought to an adjacent room where the participants will watch a brief nature video (there are two versions of this video that will be counterbalanced). After the nature video, the participants will provide ratings of awe, their feelings of connectedness to nature, and their affect using the D-FAW. Finally, participants will be asked to rate the strength of their subjective high, good drug effects, and liking of the drug effects on an iPad. The EEG headband and Embrace wristband will then be removed.

Sobering and Debriefing: Participants will then sit and play video games and/or watch TV or read until it has been a total of 4 hours since their vape session ended, and the participants report feeling completely sober. The room is equipped with couches, chairs, a TV with streaming platforms, and a video game system. Snacks (e.g., fruit snacks, granola bars, hot pockets, uncrustables, chips, chocolate bars, nuts, jerky, soda, juice, chocolate milk, water) will also be available for participants to consume while they wait. This room is equipped with a two-way mirror, and an RA will monitor participants via the window in the adjacent room to ensure the participants do not attempt to leave the lab and to monitor and record the snacks/beverages participants choose to consume and the activities the participants choose to engage in while the participants sober up. Participants will be informed that the RA is in the adjoining room, monitoring them, and that the participants can call them for assistance at any time. The RA will enter the room every 30 minutes to collect intoxication ratings. Participants will also be asked to rate how much they enjoyed each food product or beverage they consumed in the prior 30 minutes using a 0 (dislike very much) to 10 (like very much) rating scale. Participants will be debriefed after it has been a total of 4 hours have passed since their vape session ended, and they report feeling sober (give a 0 on the intoxication rating scale).

Participants will then return for their second session, which will be identical to the first, except those administered 20 mg of THC in session 1 will be administered placebo in session 2, and those administered placebo in session 2 will be administered 20 mg of THC in session 2. Participants will be debriefed at the end of session 2.

ELIGIBILITY:
Inclusion Criteria:

* be 21 years of age or older
* be fluent in English
* use of cannabis at least once a week for at least one year
* inhalation as their typical method of administration
* be willing to abstain from cannabis on the day of their scheduled testing session

Exclusion Criteria:

* neurological conditions (e.g., neurodegenerative disorders, severe head injury, multiple concussions)
* serious psychiatric conditions (e.g., psychosis, bipolar disorder)
* family history of psychosis
* intellectual disabilities or learning disorders (e.g., dyslexia)
* chronic medical conditions that affect cognition or increase risk of cannabis use or exposure to cold water (e.g., heart disease, diabetes, Reynaud's disease, history of frostbite, peripheral neuropathy, history of fainting or seizures, fractures or wounds on both hands or wrists),
* heart disease
* BMI > 34
* pregnant or lactating
* use of illicit drugs in past 6 months
* heavy use of alcohol (drinking >4 drinks >4 times per week)
* nicotine/tobacco use
* have experienced a severe adverse reaction to cannabis (e.g., panic attack, psychosis)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Event-Based Prospective Memory - Number of Difficulty Ratings Provided | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Event-based prospective memory will be assessed using a difficulty ratings task. At the beginning of the session, participants will be asked to try to remember to rate how difficult they found each test immediately after it is completed, using a 0 (not at all difficult) to 10 (extremely difficult) scale. The primary outcome of interest is the number of difficulty ratings they remember to provide.
Time-Based Prospective Memory - Token Task | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Time-based prospective memory will be assessed using a token task. Participants will be instructed to try to remember to request a token every 10 minutes. A clock will be positioned face down on the table for them to refer to the time, and we will record their clock-checking behavior. The primary outcome is the number of times they remember to request the token, out of the total time of the cognitive assessment session.
Cognitive Flexibility - N-back Test Accuracy | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Cognitive flexibility and working memory updating will be assessed using the N-back test. Participants are shown strings of letters one at a time and are instructed to indicate whenever a letter appears that matches the letter shown two trials earlier. Outcomes include the percentage of correct responses made (i.e., the number of times they correctly recognize that the current letter matches the one from two trials before, etc.).
Cognitive Flexibility - N-back Reaction Time | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Cognitive flexibility and working memory updating will be assessed using the N-back test. Participants are shown strings of letters one at a time and are instructed to indicate whenever a letter appears that matches the letter shown two trials earlier. Outcomes include the mean reaction time (milliseconds) for correct responses on the task.
Cognitive Flexibility - N-back ERP | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Cognitive flexibility and working memory updating will be assessed using the N-back test. Participants are shown strings of letters one at a time and are instructed to indicate whenever a letter appears that matches the letter shown two trials earlier. The Muse S Athena wearable EEG device will capture time-locked event-related potential data during this task.
Verbal Working Memory - Digit Span Backwards | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Verbal working memory will be assessed using the Backwards portion of the Digit Span Test. For this test, participants are read lists of digits (of increasing lengths) and are asked to recall them in reverse order. The primary outcome of interest is the total number of correct trials.
Planning - Tower Test Total Achievement Score | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Planning and problem-solving abilities will be assessed using the Tower Test. Participants are asked to move disks to reach a specified end configuration in as few moves as possible. They can move only one disk at a time and cannot place a larger disk on top of a smaller disk. Outcomes on this task include the Total Achievement Score across the tower problems, which reflects planning effectiveness.
Planning - Tower Test Rule Violations | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Planning and problem-solving abilities will be assessed using the Tower Test. Participants are asked to move disks to reach a specified end configuration in as few moves as possible. They can move only one disk at a time and cannot place a larger disk on top of a smaller disk. Outcomes on this task include the number of rule violations (e.g., moving stacking a larger disk on top of a smaller one).
Planning - Zoo Maps Test Total Achieved Score | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Planning and strategic thinking will be assessed using the Zoo Maps Test. Participants must plan a route through a provided zoo map while adhering to specified rules and efficiency constraints. For example, they may be instructed to start at the entrance, end at the picnic area, and use the designated paths only once. Outcomes on this task include the total achieved score, representing accuracy when generating a self-directed route under the provided constraints.
Planning - Zoo Maps Test Rule Violations | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Planning and strategic thinking will be assessed using the Zoo Maps Test. Participants must plan a route through a provided zoo map while adhering to specified rules and efficiency constraints. For example, they may be instructed to start at the entrance, end at the picnic area, and use the designated paths only once. Outcomes on this task include the number of rule violations on the task.
Inhibitory Control - Stroop Test Interference Score | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Inhibitory control will be assessed using the Stroop test. Participants will be shown words whose letters are in a specific color (e.g., the word "blue" in red letters. They will be tasked with naming the color of the word, which may be incongruent with the word itself. Outcomes on this task include the interference score, which reflects the difference in reaction times between the incongruent and congruent trials.
Inhibitory Control - Stroop Test Accuracy | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Inhibitory control will be assessed using the Stroop test. Participants will be shown words whose letters are in a specific color (e.g., the word "blue" in red letters. They will be tasked with naming the color of the word, which may be incongruent with the word itself. Outcomes on this task include the percentage of correct responses on incongruent trials.
Inhibitory Control - Stroop Test ERP | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Inhibitory control will be assessed using the Stroop test. Participants will be shown words whose letters are in a specific color (e.g., the word "blue" in red letters. They will be tasked with naming the color of the word, which may be incongruent with the word itself. The Muse S Athena wearable EEG device will capture time-locked event-related potential data during this task.
Inhibitory Control - Flanker Test Interference Score | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Inhibitory control and attention will be assessed using the Flanker Test. Participants will respond to a central target stimulus (e.g., an arrow pointing in one direction) while ignoring surrounding distractor stimuli, that may be either congruent (e.g., an arrow pointing the same way) or incongruent (e.g., an arrow pointing the opposite way). Outcomes on this task include the interference score, which is the difference in reaction time between incongruent and congruent trials.
Inhibitory Control - Flanker Test Accuracy | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Inhibitory control and attention will be assessed using the Flanker Test. Participants will respond to a central target stimulus (e.g., an arrow pointing in one direction) while ignoring surrounding distractor stimuli, that may be either congruent (e.g., an arrow pointing the same way) or incongruent (e.g., an arrow pointing the opposite way). Outcomes on this task include the percentage of correct responses across trial types.
Inhibitory Control - Flanker Test ERP | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Inhibitory control and attention will be assessed using the Flanker Test. Participants will respond to a central target stimulus (e.g., an arrow pointing in one direction) while ignoring surrounding distractor stimuli, that may be either congruent (e.g., an arrow pointing the same way) or incongruent (e.g., an arrow pointing the opposite way). The Muse S Athena wearable EEG device will capture time-locked event-related potential data during this task.
Cognitive Control - Oddball Task Target Detection Accuracy | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Cognitive control and sustained attention will be assessed using the Oddball Task. Participants will be asked to tap the screen when they see an infrequent red ball stimulus, and refrain from tapping when they see a green ball stimulus. Outcomes include the percentage of correctly identified target stimuli.
Cognitive Control - Oddball Task Target Reaction Time | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Cognitive control and sustained attention will be assessed using the Oddball Task. Participants will be asked to tap the screen when they see an infrequent red ball stimulus, and refrain from tapping when they see a green ball stimulus. Outcomes include the mean reaction time (milliseconds) for responses to target stimuli.
Cognitive Control - Oddball Task ERP | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Cognitive control and sustained attention will be assessed using the Oddball Task. Participants will be asked to tap the screen when they see an infrequent red ball stimulus, and refrain from tapping when they see a green ball stimulus. The Muse S Athena wearable EEG device will capture time-locked event-related potential data during this task.
Cognitive Flexibility - Wisconsin Card Sorting Test Perseverative Errors | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Cognitive flexibility (attentional set-shifting) will be assessed using the Wisconsin Card Sorting Task (WCST). Participants will sort cards of various shapes, colors, and numbers to match an undisclosed rule. After each card placement, participants will receive either "correct" or "incorrect" feedback to help them deduce the sorting rule. The sorting rule will periodically and unpredictably change (typically after a series of correct responses), and the participant must then infer the new rule. Outcomes on this task include the number of perseverative errors (i.e., failure to switch sorting strategies when the old sorting rule becomes incorrect).
Cognitive Flexibility - Wisconsin Card Sorting Test Categories Completed | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Cognitive flexibility (attentional set-shifting) will be assessed using the Wisconsin Card Sorting Task (WCST). Participants will sort cards of various shapes, colors, and numbers to match an undisclosed rule. After each card placement, participants will receive either "correct" or "incorrect" feedback to help them deduce the sorting rule. The sorting rule will periodically and unpredictably change (typically after a series of correct responses), and the participant must then infer the new rule. Outcomes on this task include the total number of sorting categories correctly completed.
Cognitive Flexibility - Wisconsin Card Sorting Test Failure-to-Maintain-Set Errors | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Cognitive flexibility (attentional set-shifting) will be assessed using the Wisconsin Card Sorting Task (WCST). Participants will sort cards of various shapes, colors, and numbers to match an undisclosed rule. After each card placement, participants will receive either "correct" or "incorrect" feedback to help them deduce the sorting rule. The sorting rule will periodically and unpredictably change (typically after a series of correct responses), and the participant must then infer the new rule. Outcomes on this task include the number of errors reflecting a breakdown in sustained performance (e.g., not following the correct sorting rule after having learned it and without feedback indicating the rule has changed).
Cognitive Flexibility - Verbal Fluency, Category Switching Fluency | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Cognitive flexibility (category switching) will be assessed using the verbal fluency category switching task. Participants will be given two categories (e.g., fruits and furniture) and be asked to generate words that belong to those categories, in alternating order, within a time limit of 60 seconds. Outcomes on this task include the category fluency score, which is the number of correct words generated.
Cognitive Flexibility - Verbal Fluency, Category Switching Accuracy | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Cognitive flexibility (category switching) will be assessed using the verbal fluency category switching task. Participants will be given two categories (e.g., fruits and furniture) and be asked to generate words that belong to those categories, in alternating order, within a time limit of 60 seconds. Outcomes on this task include category switching accuracy, which is the number of correct switches between the categories.
Stressor Challenge - Maastricht Acute Stress Test Subjective Pain Ratings | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Participants will complete an acute stress challenge, involving alternating trials of a physical stressor (placing their hand in a cooler of cold water) and a cognitive stressor (mental arithmetic). Outcomes on this test include subjective pain ratings, which are collected after each cold water trial on a 0 (not at all painful) to 10 (extremely painful) scale.
Stressor Challenge - Maastricht Acute Stress Test Subjective Stress Ratings | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Participants will complete an acute stress challenge, involving alternating trials of a physical stressor (placing their hand in a cooler of cold water) and a cognitive stressor (mental arithmetic). Outcomes on this test include subjective stress ratings, which are collected after each mental math trial on a 0 (not at all stressed) to 10 (extremely stressed) scale.
EEG Power | This outcome will be continuously assessed during both sessions, from baseline (i.e., during the testing session but before treatment) through two hours post-treatment.
  The Muse S Athena wearable EEG device will be worn by participants for the duration of the session, up until they are left to relax and sober up at the end of the session. The EEG device will be continuously recording, to allow for later quantification of power (e.g., theta, gamma, etc.) using spectral density analysis.
Awe Ratings | This outcome will be assessed during both sessions, within two hours post-treatment.
  Participants will complete ratings of awe after watching a brief (~20 minute) nature video.
Connectedness to Nature Ratings | This outcome will be assessed during both sessions, within two hours post-treatment.
  Participants will complete ratings of their feelings of connectedness to nature after watching a brief (~20 minute) nature video.

SECONDARY OUTCOMES:
Event-Based Prospective Memory - Difficulty Ratings | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Event-based prospective memory will be assessed using a difficulty ratings task. At the beginning of the session, participants will be asked to try to remember to rate how difficult they found each test immediately after it is completed, using a 0 (not at all difficult) to 10 (extremely difficult) scale. The primary outcome of interest is the self-reported difficulty of each task completed.
Time-Based Prospective Memory - Token Task Clock-Checking | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Time-based prospective memory will be assessed using a token task. Participants will be instructed to try to remember to request a token every 10 minutes. A clock will be positioned face down on the table for them to refer to the time, and we will record their clock-checking behavior. The primary outcome is the number of times they check the clock over the duration of the cognitive assessment session.
Planning - Tower Test Time to Completion | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Planning and problem-solving abilities will be assessed using the Tower Test. Participants are asked to move disks to reach a specified end configuration in as few moves as possible. They can move only one disk at a time and cannot place a larger disk on top of a smaller disk. Outcomes on this task include the time taken to complete each tower problem.
Cogntiive Flexibility - Verbal Fluency, Category Switching Errors | This outcome will be assessed during both sessions, within 90 minutes post-treatment.
  Cognitive flexibility (category switching) will be assessed using the verbal fluency category switching task. Participants will be given two categories (e.g., fruits and furniture) and be asked to generate words that belong to those categories, in alternating order, within a time limit of 60s. Outcomes on this task include repetition and intrusion (i.e., non-category words) errors.
Baseline (T0) Intoxication Rating | This outcome will be assessed during both sessions at baseline (i.e., during the testing session but before treatment).
  Participants will be asked to rate how high they feel using a scale from 0 (not high at all) to 10 (extremely high) prior to completing any study tasks.
Post-Treatment (T1) Intoxication Rating | This outcome will be assessed during both sessions immediately after their vaping session.
  Participants will be asked to rate how high they feel using a scale from 0 (not high at all) to 10 (extremely high) immediately after their vaping session.
Post-Treatment (T1) Good Drug Effects Rating | This outcome will be assessed during both sessions immediately after their vaping session.
  Participants will be asked to rate the level of good drug effects they are experiencing using a scale from 0 (none) to 10 (a lot) immediately after their vaping session.
Post-Treatment (T1) Drug Effects Liking Rating | This outcome will be assessed during both sessions immediately after their vaping session.
  Participants will be asked to rate how much they like the drug effects they are experiencing using a scale from 0 (not at all) to 10 (a lot) immediately after their vaping session.
Post-Stress Challenge (T2) Intoxication Rating | This outcome will be assessed during both sessions immediately after the stress challenge.
  Participants will be asked to rate how high they feel using a scale from 0 (not high at all) to 10 (extremely high) immediately after the stress challenge.
Post-Stress Challenge (T2) Good Drug Effects Rating | This outcome will be assessed during both sessions immediately after the stress challenge.
  Participants will be asked to rate the level of good drug effects they are experiencing using a scale from 0 (none) to 10 (a lot) immediately after the stress challenge.
Post-Stress Challenge (T2) Drug Effects Liking Rating | This outcome will be assessed during both sessions immediately after the stress challenge.
  Participants will be asked to rate how much they like the drug effects they are experiencing using a scale from 0 (not at all) to 10 (a lot) immediately after the stress challenge.
Post-Nature Video (T3) Intoxication Rating | This outcome will be assessed during both sessions immediately after the nature video.
  Participants will be asked to rate how high they feel using a scale from 0 (not high at all) to 10 (extremely high) immediately after the nature video.
Post-Nature Video (T3) Good Drug Effects Rating | This outcome will be assessed during both sessions immediately after the nature video.
  Participants will be asked to rate the level of good drug effects they are experiencing using a scale from 0 (none) to 10 (a lot) immediately after the nature video.
Post-Nature Video (T3) Drug Effects Liking Rating | This outcome will be assessed during both sessions immediately after the nature video.
  Participants will be asked to rate how much they like the drug effects they are experiencing using a scale from 0 (not at all) to 10 (a lot) immediately after the nature video.
Cortisol Change Score: Baseline to Post-Treatment | This outcome will be computed from measures collected at baseline (i.e., during the testing session but before treatment) and immediately after treatment.
  The change in salivary cortisol concentrations will be calculated between baseline and post-treatment (THC or placebo) assessments.
Cortisol Change Score: Baseline to Post-Cognitive Assessment | This outcome will be computed from measures collected at baseline (i.e., during the testing session but before treatment) and immediately after cognitive assessments.
  The change in salivary cortisol concentrations will be calculated between baseline and post-cognitive session assessments.
Cortisol Change Score: Baseline to Post-Stress Challenge | This outcome will be computed from measures collected at baseline (i.e., during the testing session but before treatment) and immediately after the stress challenge.
  The change in salivary cortisol concentrations will be calculated between baseline and post-cognitive session assessments.
Cortisol Change Score: Post-Cognitive Assessment to Post-Stress Challenge | This outcome will be computed from measures collected immediately following the cognitive assessment session and immediately after the stress challenge.
  The change in salivary cortisol concentrations will be calculated between post-cognitive assessment and post-stress challenge assessments.
Affect Change Score: Baseline to Post-Treatment | This outcome will be computed from measures collected at baseline (i.e., during the testing session but before treatment) and immediately after treatment.
  The change in affect, assessed using the Daniels Five-Factor Measure of Affective Well-Being, will be calculated between baseline and post-treatment (THC or placebo) assessments.
Affect Change Score: Baseline to Post-Cognitive Assessment | This outcome will be computed from measures collected at baseline (i.e., during the testing session but before treatment) and immediately after cognitive assessments.
  The change in affect, assessed using the Daniels Five-Factor Measure of Affective Well-Being, will be calculated between baseline and post-cognitive session assessments.
Affect Change Score: Baseline to Post-Stress Challenge | This outcome will be computed from measures collected at baseline (i.e., during the testing session but before treatment) and immediately after the stress challenge.
  The change in affect, assessed using the Daniels Five-Factor Measure of Affective Well-Being, will be calculated between baseline and post-stress challenge assessments.
Affect Change Score: Post-Cognitive Assessment to Post-Stress Challenge | This outcome will be computed from measures collected immediately following the cognitive assessment session and immediately after the stress challenge.
  The change in affect, assessed using the Daniels Five-Factor Measure of Affective Well-Being, will be calculated between post-cognitive assessment and post-stress challenge assessments.
Affect Change Score: Baseline to Post-Nature Video | This outcome will be computed from measures collected at baseline (i.e., during the testing session but before treatment) and immediately after the nature video.
  The change in affect, assessed using the Daniels Five-Factor Measure of Affective Well-Being, will be calculated between baseline and post-nature video assessments.
Affect Change Score: Post-Stress Challenge to Post-Nature Video | This outcome will be computed from measures collected immediately following the stress challenge and immediately following the nature video.
  The change in affect, assessed using the Daniels Five-Factor Measure of Affective Well-Being, will be calculated between post-stress challenge and post-nature video assessments.

OTHER OUTCOMES:
Cannabis Consumption Patterns | This outcome will be assessed at baseline (i.e., during the testing session but before treatment).
  As part of their baseline assessments, participants will complete the Daily Sessions, Frequency, Age of Onset, and Quantity of Cannabis Use Inventory, which is a standardized, valid, and reliable measure of their cannabis consumption patterns. The information from this survey will be used to characterize the sample and determine cannabis use-related covariates that should be controlled for in analyses.
Drug Screen | This outcome will be assessed during both sessions at baseline (i.e., during the testing session but before treatment).
  Participants will complete a 12-panel urine drug test to ensure they test positive for cannabis/THC but no other illicit drugs.
Electrodermal Activity | This outcome will be continuously assessed during both sessions from before drug/placebo administration to immediately before they leave the lab (approximately 5 hours).
  An Empatica E4 medical-grade device will be used to collect continuous measures of electrodermal activity.
Heart Rate/Heart Rate Variability | This outcome will be continuously assessed during both sessions from before drug/placebo administration to immediately before they leave the lab (approximately 5 hours).
  An Empatica E4 medical-grade device will be used to collect continuous measures of heart rate/heart rate variability.
Temperature | This outcome will be continuously assessed during both sessions from before drug/placebo administration to immediately before they leave the lab (approximately 5 hours).
  An Empatica E4 medical-grade device will be used to collect continuous measures of temperature.
Motion | This outcome will be continuously assessed during both sessions from before drug/placebo administration to immediately before they leave the lab (approximately 5 hours).
  An Empatica E4 medical-grade device will be used to collect continuous measures of motion.
Post-Session Intoxication Ratings | This outcome will be assessed every 30 minutes from 2 hours post-dose through 4 hours post-dose (or until the participant reports sobriety, whichever occurs later).
  Participants will be asked to rate how high they feel using a scale from 0 (not high at all) to 10 (extremely high) while relaxing and sobering up, following the rest of their session.
Verbal Intelligence (IQ) | This outcome will be assessed at baseline (i.e., during the testing session but before treatment).
  As part of their baseline assessments, participants will complete the Wechsler Test of Adult Reading as an index of verbal IQ. This will provide a metric to ensure that participants are equivalent (i.e., statistically comparable) in verbal IQ. This test simply requires participants to pronounce a list of words (e.g., treaties, knead, liaison). The outcome of interest is the total number of correctly pronounced words.
Depression - Center for Epidemiologic Studies Depression Scale | This outcome will be assessed at baseline (i.e., during the testing session but before treatment).
  As part of their baseline assessments, participants will complete the Center for Epidemiologic Studies Depression Scale. Higher scores indicate more frequent and more severe depressive symptoms. Potential scores range from 0-60. The information from this survey will be used to characterize the sample and determine potential covariates that should be controlled for in analyses.
Anxiety - Beck Anxiety Inventory | This outcome will be assessed at baseline (i.e., during the testing session but before treatment).
  As part of their baseline assessments, participants will complete the Beck Anxiety Inventory. Higher scores indicate greater anxiety severity. Potential scores range from 0-63. The information from this survey will be used to characterize the sample and determine potential covariates that should be controlled for in analyses.
ADHD Symptoms - Barkley Adult ADHD Rating Scale - IV | This outcome will be assessed at baseline (i.e., during the testing session but before treatment).
  As part of their baseline assessments, participants will complete the Barkley Adult ADHD Rating Scale (IV). Higher scores indicate greater ADHD symptom frequency and severity. Potential scores range from 0-54. The information from this survey will be used to characterize the sample and determine potential covariates that should be controlled for in analyses.
Emotion Regulation - Difficulties in Emotion Regulation Scale | This outcome will be assessed at baseline (i.e., during the testing session but before treatment).
  As part of their baseline assessments, participants will complete the Difficulties in Emotion Regulation Scale. Higher scores indicate greater difficulties with emotion regulation across domains. Potential scores range from 36-180. The information from this survey will be used to characterize the sample and determine potential covariates that should be controlled for in analyses.
Vaping Session - Total Puffs | This outcome will be assessed during the vaping session (i.e., from the beginning of the vaping session until the end of the vaping session) during both sessions. This vaping session will occur immediately after the baseline assessments.
  The principal investigator supervising the vaping session will record the total number of puffs the participant inhales.
Vaping Session - Inhalation/Hold Duration | This outcome will be assessed during the vaping session (i.e., from the beginning of the vaping session until the end of the vaping session) during both sessions. This vaping session will occur immediately after the baseline assessments.
  The principal investigator supervising the vaping session will record the duration of the participant's inhalations and holds during the vaping session.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J McLaughlin, PhD, Principal Investigator — Washington State University; Carrie Cuttler, PhD, Principal Investigator — Washington State University
Locations (1):
- Washington State University, Pullman, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon request and after publication of our primary findings.
Supporting Information: Study Protocol, ICF
Time Frame: After the publication of primary findings.
Access Criteria: The IPD will be available upon email request to one of the PIs on this study. De-identified data and the study protocol, statistical analysis plan, and informed consent form can/will be shared upon request.